CLINICAL TRIAL: NCT06014073
Title: A Phase 1/2 Single-center Study Evaluating the Safety and Efficacy of TRAC and Power3 (SPPL3) Genes Knock-out Allogeneic CD19-targeting CAR-T Cell (ATHENA) Therapy in Adults With Refractory/Relapsed B-cell Non-Hodgkin Lymphoma
Brief Title: TRAC and Power3 (SPPL3) Genes Knock-out Allogeneic CD19-targeting CAR-T Cell Therapy in r/r B-NHL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Peking University (Other); EdiGene Inc. (Industry)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-082
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Non Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with refractory or relapsed B-cell NHL (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, TRAC and Power3 (SPPL3) Gene Knock-out Allogeneic CD19-targeting CAR-T.
  Interventions: Biological: TRAC and Power3 (SPPL3) Genes Knock-out Allogeneic CD19-targeting CAR-T cell (ATHENA CAR-T); Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: TRAC and Power3 (SPPL3) Genes Knock-out Allogeneic CD19-targeting CAR-T cell (ATHENA CAR-T) — Phase 1 dose escalation (3+3) : dose 1 (1 × 10^6 cells/kg) , dose 2 (3 × 10^6 cells/kg), dose 3 (1 × 10^7 cells/kg); Phase 2 : dose of RP2D.
  No more than 2 × 10^5 per kilogram of allogenic residual CD3+T cells harbouring in grafts can only be released for recipient infusion.
Drug: Fludarabine — Intravenous fludarabine 30~50 mg/m^2/day on days -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 500~1000 mg/m^2/day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
ATHENA chimeric antigen receptor (CAR)-T, a CD19-directed CAR-T cell immunotherapy comprised of allogeneic T cells prepared for the treatment of relapsed or refractory (r/r) B-cell non-Hodgkin's lymphoma (NHL). The cells are from healthy adult volunteer donors that are knocked out of TRAC and Power3 (SPPL3) genes ex vivo using CRISPR-Cas9 gene editing components. In this study, a second-generation anti-CD19 CAR prototype was constructed, bearing murine FMC63 single-chain variant fragment (scFv) together with intracellular CD28 co-stimulatory and CD3ζ signaling domains linked by a CD28 sequence comprising the hinge and transmembrane domains.

This is a single center, prospective, open-label, single-arm, phase 1/2 study. A total of around 30 patients with r/r B-cell NHL will be enrolled in the study and receive allogeneic CD19-CAR-T cell infusion. Phase 1 (n=6 to 18) is a dose escalation part, and phase 2 (n=10 to 12) is a expansion cohort part. The primary objective of this study was to evaluate the safety and efficacy of ATHENA CAR-T cell therapy in patients with r/r B-cell NHL.

DETAILED DESCRIPTION:
Phase 1 (dose escalation)

In phase 1, 6-18 subjects will be enrolled. Subjects will receive 3 doses of ATHENA CAR-T cell therapy ( 1× 10^6 cells/kg、3× 10^6 cells/kg、1 × 10^7 cells/kg) increases from low dose to high dose according to the "3 + 3" principle:

Three (3) subjects are enrolled in a cohort corresponding to a dose level. If 1 subject in a cohort of 3 subjects experiences a dose-limiting toxicity (DLT), 3 additional subjects will be enrolled at the current dose level. For safety purposes, the administration of ATHENA CAR T will be staggered by 28 days between the first two subjects in each cohort. And for each of the remaining cohorts, the administration of ATHENA CAR-T will be staggered by 28 days before enter into the next cohort.

Phase 2 (expansion cohort)

In phase 2, 10 to 12 subjects will be enrolled and receive ATHENA CAR-T cell infusion at dose of recommended phase 2 dose (RP2D), which will be determined based on the maximum tolerated dose (MTD), occurrence of DLT, the obtained efficacy results, pharmacokinetics/pharmacodynamics and other data according to the phase 1.

Objectives

The primary objectives of the phase 1 were to evaluate the tolerability and safety of ATHENA CAR-T in patients with r/r B-cell NHL, and determine RP2D. The primary purpose of the phase 2 study was to evaluate the efficacy of ATHENA CAR-T in the above population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 (inclusive).
2. Subjects who meet the following requirements:

   2.1 Histologically confirmed refractory/relapsed B cell NHL, including the following types defined by WHO 2016:
   * Diffuse large B-cell lymphoma (DLBCL) not otherwise specified;
   * Primary mediastinal (thymic) large B-cell lymphoma (PMBCL);
   * Transformed follicular lymphoma (TFL);
   * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (HGBCL);
   * Follicular lymphoma (FL);
   * Mantle cell lymphoma (MCL) (pathologically confirmed, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1);
   * Marginal zone lymphoma (MZL), including nodal or splenic marginal zone B-cell lymphoma and mucosa-associated lymphoid tissue (MALT) lymphoma.

   2.2 Relapsed disease is defined as disease progression (PD) after achieving disease remission (including CR and PR) with the latest standard regimen.

   2.3 Refractory disease is defined as no CR to first-line therapy:
   * Evaluation of PD (never reached response or SD) after standard first-line treatment, or
   * SD as best response after at least 4 cycles of first-line therapy (eg,4 cycles of R-CHOP), or
   * PR as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 6 months of therapy, or
   * Refractory post-autologous stem cell transplant (ASCT) i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals) ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy.

   2.4 Individuals who are intolerant to standard treatment can also be included in the study in the investigator's judgment.
3. Individuals must have received adequate prior therapy:

   3.1 For MCL, prior therapy must have included:
   * Anthracycline or bendamustine-containing chemotherapy and
   * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
   * Bruton's tyrosine kinase inhibitor (BTKi).

   3.2 For other types, prior therapy must have included:
   * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
   * Anthracycline containing chemotherapy regimen.

   3.3 For individual with transformed FL must have relapse or refractory disease after transformation to DLBCL.
4. At least 1 measurable lesion: lymph node site with a long axis >1.5cm, extranodal site with a long axis >1.0cm (according to Lugano2014). Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
5. CD19 positive (detected by immunohistochemistry [IHC]).
6. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for hematological toxicities and clinically non-significant toxicities such as alopecia).
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
8. Absolute neutrophil count (ANC) ≥ 1 x 10^9/L, Platelet count ≥50 x 10^9/L, hemoglobin (Hgb) ≥ 80g/L (hemocytopenia caused by lymphoma invasion of bone marrow is not subject to conditions above).
9. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   9.1 Serum creatinine≤1.5 upper limit of normal (ULN) or creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min.

   9.2 Serum alanine aminotransferase / aspartate aminotransferase (ALT/AST) ≤ 3 upper limit of normal (ULN); Total bilirubin ≤ 1.5 ULN, except in subjects with 3) Gilbert's syndrome.

   9.3 Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings.

   9.4 Coagulation Function: International Normalized Ratio (INR) ≤ 1.5 times the upper limit of normal (ULN), and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN.

   9.5 Baseline oxygen saturation >91% on room air.
10. Subjects of both genders who are willing to practice birth control from the time of consent through 6 months after the completion of conditioning chemotherapy. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential).
11. Voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Expected survival time < 3 months per Principal Investigator's opinion.
2. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years.
3. Autologous stem cell transplant with therapeutic intent within 3 months of planned ATHENA CAR-T infusion.
4. History of allogeneic stem cell transplantation.
5. Prior CD19 targeted therapy.
6. Patients who have used any of the following agents or treatments within a specific period of time:

   6.1 Received any chemotherapy drugs or small molecule targeted drugs within 2 weeks prior to lymphodepletion;

   6.2 Received any monoclonal antibodies, antibody drug conjugates (ADCs), or bispecific antibodies within 3 weeks prior to lymphodepletion;

   6.3 Received radiotherapy within 6 weeks prior to lymphodepletion. However, if disease progressed at the site of radiotherapy, or if there are positive lesions detected by PET-CT at non-radiotherapy sites, enrollment is allowed.
7. Prior CAR-T therapy or other genetically modified T cell therapy.
8. Subjects with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of central nervous system (CNS) lymphoma or primary CNS lymphoma.
9. History of severe, immediate hypersensitivity reaction attributed to lymphodepletion drugs or any component of ATHENA CAR-T.
10. Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management.
11. Uncontrolled or active infectious diseases, such as human immunodeficiency virus (HIV) infection, acute or chronic active hepatitis B or C, epstein-barr virus (EBV), and cytomegalovirus (CMV) infection.
12. History or presence of central nervous system (CNS) disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
13. Subjects with cardiac atrial or cardiac ventricular lymphoma involvement.
14. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
15. Expected or possible requirement for urgent therapy within 6 weeks due to ongoing or impending oncologic emergency (eg, tumor mass effect, tumor lysis syndrome).
16. Primary immunodeficiency.
17. History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
18. History of symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within 6 months of enrollment.
19. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment.
20. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
21. Vaccine ≤ 6 weeks prior to planned start of conditioning regimen.
22. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of adverse events (AE) defined as DLT | First infusion date of CAR-T cells up to 28 days
  DLT is defined as any AE related to the investigational drug that occurs within 28 days after administration of the ATHENA CAR-T and meets any one of the criteria listed in the DLT criteria. The severity of AE will be assessed according to NCI-CTCAE v5.0. cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) will be evaluated according to the standards released by ASTCT in 2019. Graft-versus-host-disease(GvHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium.
  * Grade 3 aGVHD that does not resolve to Grade 1 or 2 within 7 days, with the exception of isolated skin involvement aGVHD;
  * Grade 4 CRS or grade 3 CRS that does not resolve to grade 2 or lower within 2 weeks;
  * Grade 3 ICANS lasting for ≥7 days or Grade 4 ICANS;
  * Any other Grade ≥4 and Grade 3 AE related to the ATHENA CAR-T that lasts for ≥14 days, except hematology toxicity.
Phase 1: RP2D | 12 months
  The RP2D was determined through phase 1 study.
Phase 2: 3-month objective response rate (ORR) | 3 months
  ORR is defined as the proportion of patients who have achieved complete response (CR) and partial response (PR) assessed by investigators and based on the Lugano 2014 assessment criterion.
Phase 2: CR rate | 24 months
  CR rate is defined as the proportion of patients who have achieved CR assessed by investigators and based on the Lugano 2014 assessment criterion.
Phase 2: Duration of Response (DOR) | 24 months
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators and based on the Lugano 2014 assessment criterion for r/r B-cell NHL, or death regardless of cause.
Phase 2: Overall Survival (OS) | 24 months
  OS is defined as the time from CAR-T cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Phase 2: Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from the CAR-T cells infusion date to the date of disease progression assessed by investigators and based on the Lugano 2014 assessment criterion, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.

SECONDARY OUTCOMES:
Phase 1 and phase 2: Pharmacokinetics: Levels of ATHENA CAR-positive T cells circulating in blood over time | 12 months
  Number and copy number of ATHENA CAR-T cells were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (until CAR-T cells were not detected for two consecutive times) to detect the number and copy number of CAR-T cells, and to evaluate the pharmacokinetics of CAR-T.
Phase 1 and phase 2: Pharmacodynamics: Levels of CD19+ cells and serum cytokines in peripheral blood | Up to 28 days after infusion
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP), ferritin.
Phase 1: 3-month ORR | 3 months
  ORR is defined as the proportion of patients who have achieved CR and PR assessed by investigators and based on the Lugano 2014 assessment criterion.
Phase 1: OS | 24 months
  The definition of OS has already been mentioned above
Phase 1: PFS | 24 months
  The definition of PFS has already been mentioned above
Phase 2: Incidence of AE and clinical significant changes in safety lab values | 24 months
  AE is defined as any adverse medical event from the date of enrollment to 24 months after CAR-T cells infusion.

OTHER OUTCOMES:
Phase 1: Levels of donor-specific antibody (DSA) in blood. | 12 months
  DSA refers to the specific antibody produced in the recipient's body targeting donor antigens after receiving CAR-T cell infusion from healthy donors.
Phase 1: Levels of human anti-mouse antibodies (HAMA) | 12 months
  The levels of human against murine scFv antibodies in blood

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (3):
- China (3):
  - Biotherapeutic Department, Chinese PLA General Hospital, Beijing
  - EdiGene Inc, Beijing
  - School of Life Sciences, Peking University, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu Z, Shi J, Lamao Q, Qiu Y, Yang J, Liu Y, Liang F, Sun X, Tang W, Chen C, Yang Q, Wang C, Li Z, Zhang H, Yang Z, Zhang Y, Yi Y, Zheng X, Sun Y, Ma K, Yu L, Yang H, Wang Z, Zheng W, Yang L, Zhang Z, Zhang Y, Wu Z, Wang Y, Wong CCL, Jin M, Yuan P, Han W, Wei W. Glycan shielding enables TCR-sufficient allogeneic CAR-T therapy. Cell. 2025 Oct 30;188(22):6317-6334.e21. doi: 10.1016/j.cell.2025.07.046. Epub 2025 Aug 21. PMID 40845838